CLINICAL TRIAL: NCT06861374
Title: Bivalirudin Plus High-Dose Infusion Versus Heparin Monotherapy in Patients with ST-Segment Elevation Myocardial Infarction Undergoing Percutaneous Coronary Intervention After Fibrinolysis: a Randomized Trial
Brief Title: Bivalirudin with Prolonged Infusion During PCI Versus Heparin After Fibrinolytic Therapy
Acronym: BRIGHT-FIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF2024LSYY-321
Record Dates: First submitted 2025-03-03; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: STEMI, PCI, fibrinolysis, bivalirudin, heparin, bleeding, mortality
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Hemorrhage | interventions — bivalirudin; Heparin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bivalirudin (Experimental): bivalirudin with a prolonged infusion
  Interventions: Drug: Bivalirudin
- Heparin (Active Comparator): Heparin alone during PCI
  Interventions: Drug: Unfractionated heparin

INTERVENTIONS:
Drug: Bivalirudin — For rescued PCI, do not recommend to include patient who's ACT is more than 350s.
  If fibrinolysis is successful, monitor ACT and wait till it's lower than 350s before randomization.
  Monitor ACT before angiography, (1) if ACT<180, bivalirudin 0.75 mg/kg intravenous bolus loading dose, and immediately followed by intravenous infusion of 1.75 mg/kg/h until 2-4 hours after PCI; (2) if 180s<ACT<225s, bivalirudin 0.5mg/kg intravenous bolus loading dose, and immediately followed by intravenous infusion of 1.75 mg/kg/h until 2-4 hours after PCI; (3) if ACT>225s, bivalirudin intravenous infusion of 1.75 mg/kg/h until 2-4 hours after PCI. (4) ACT be monitored 5 minutes after the first administration, and if ACT is <225 s, intravenous injection of 0.3 mg/kg of bivalirudin should be administered, and the ACT re-checked to ensure it is >225 seconds.
  Arms: Bivalirudin
Drug: Unfractionated heparin — (1)If ACT<180s, administer an intravenous bolus of unfractionated heparin at 70 U/kg before coronary angiography, with a maximum total dose of 6000U. (2)If 180<ACT<225s, administer an intravenous bolus of unfractionated heparin at 60 U/kg before coronary angiography, with a maximum total dose of 4000U. (3)If ACT>225s, proceed directly with PCI and maintain 225s<ACT<350s.
  Arms: Heparin

SUMMARY:
This multicenter, randomized controlled trial in China aims to enroll 2,400 patients with ST-segment elevation myocardial infarction undergoing percutaneous coronary intervention (PCI) within 24 hours post-fibrinolysis. Participants will be randomly assigned in a 1:1 ratio to receive either bivalirudin or heparin, with follow-up at 30 days and 1 year. The primary endpoint is a composite of all-cause mortality and Bleeding Academic Research Consortium (BARC) type 3 or 5 bleeding at 30 days.

DETAILED DESCRIPTION:
Bivalirudin is a direct thrombin inhibitor that exhibits a reversible and transient anticoagulant effect. Randomized trials have shown conflicting results for bivalirudin in reducing the risk of bleeding for ST-segment elevation myocardial infarction (STEMI) patients undergoing primary PCI (PPCI) compared to heparin. Recently, the BRIGHT-4 study, which assigned 6016 STEMI patients to bivalirudin with a prolonged high dose infusion or heparin during PPCI, showed bivalirudin decreased the risk of a composite endpoint of all-cause mortality and bleeding. However, few studies have focused on the safety and efficacy of bivalirudin in PCI post-fibrinolysis. We therefore aim to conduct the Bivalirudin With Prolonged Infusion During PCI Versus Heparin Following Fibrinolytic Therapy (BRIGHT-FIT) trial to examine whether bivalirudin with a high-dose infusion in PCI after fibrinolysis in superior to heparin in reducing mortality and major bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Any age
* STEMI patients received fibrinolysis therapy within 12h of symptom onset and are planned to undergo PCI within 24h of symptom onset.
* Dual antiplatelet drugs must be administrated according to guidelines before PCI (loading doses and maintenance doses of aspirin and clopidogrel or ticagrelor)
* Patients requiring staged revascularization of non-culprit vessels within 30 days may be enrolled. In such cases the same antithrombotic agents and PCI procedures must be used in the staged procedure consistent with the index procedure PCI, in particular the assigned antithrombin agent heparin vs. bivalirudin);
* The subject or legal representative has been informed of the nature of the study, understood the provisions of the protocol, was able to ensure adherence, and signed informed consent.

Exclusion Criteria:

* Not suitable for PCI;
* Mechanical complications (such as ventricular septal rupture, papillary muscle rupture with acute mitral regurgitation, etc.);
* Cardiogenic shock(Killip IV)
* Known allergy or contraindications to heparin, bivalirudin, aspirin, or both clopidogrel and ticagrelor
* Patients who underwent PCI in past 30 days
* Patients in whom the investigators consider inappropriate to participate in this study (eg, have participated in another drug/instrument study or undergoing another drug/instrument study, pregnancy).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause death or BARC type 3、5 bleeding | 30days
  BARC=Bleeding academic research consortium

SECONDARY OUTCOMES:
All cause mortality | 30days and 1year
Composite of all-cause death or BARC type 2、3、5 bleeding | 30days and 1year
  BARC=Bleeding academic research consortium
Net adverse clinical events (NACE) | 30days and 1year
  NACE is defined as a composite of MACCE or BARC type 3、5 bleeding
Major adverse cardiac and cerebral events (MACCE) | 30days and 1year
  MACCE is defined as a composite of all cause death, recurrent myocardial infarction, stroke or ischemic driven target vessel revascuarlization
Stent thrombosis | 30days
  Definite or probable stent thrombosis according to Academic Research Consortium
BARC type 3、5 bleeding | 30days
  BARC=Bleeding academic research consortium
BARC type 2、3、5 bleeding | 30days
  BARC=Bleeding academic research consortium
Thrombocytopenia | 30days
  defined as platelet counts less than 150*10^9/L after treatment

IPD SHARING:
Plan to Share IPD: No